CLINICAL TRIAL: NCT04743622
Title: Comparison of Efficacy and Ocular Surface Disease Assessment Between Monoprost and BAK-preserved Latanoprost in Glaucoma or Ocular Hypertensive Patients
Brief Title: Comparison of Efficacy and Ocular Surface Disease Assessment Between Monoprost and BAK-preserved Latanoprost
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CHA University (Other)
Collaborators: Samil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIT 2019-02-020
Record Dates: First submitted 2021-01-26; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monoprost (preservative-free latanoprost eye drop) (Experimental): latanoprost : 1 drop once a day for 12 weeks to target eyes
  Interventions: Drug: Monoprost
- Xalatan (preserved latanoprost eye drop) (Active Comparator): latanoprost : 1 drop once a day for 12 weeks to target eyes
  Interventions: Drug: Xalatan

INTERVENTIONS:
Drug: Monoprost — preservative-free latanoprost 1 drop once a day for 12 weeks to target eyes
  Other Names: Preservative-free latanoprost
  Arms: Monoprost (preservative-free latanoprost eye drop)
Drug: Xalatan — preserved latanoprost 1 drop once a day for 12 weeks to target eyes
  Other Names: Preserved latanoprost
  Arms: Xalatan (preserved latanoprost eye drop)

SUMMARY:
Comparison of Efficacy and Ocular Surface Disease Assessment Between Monoprost and BAK-preserved Latanoprost in Glaucoma or Ocular Hypertensive Patients : Phase 4, Parallel Group Design, Investigator-blind, Active-control, Randomized, Multi-center Study

DETAILED DESCRIPTION:
Not provided

ELIGIBILITY:
Inclusion Criteria:

* IOP >/= 15mmHg and < 40 mmHg in each eye using Goldmann applanation tonometry at visit 2
* Written consent voluntarily to participate in this clinical trial

Exclusion Criteria:

* Patients with closed-angle, congenital glaucoma or secondary glaucoma caused by steroid drugs, etc.
* best-corrected visual acuity 20/80 or less
* Patients who have ongoing medical history of ocular inflammation
* central corneal thickness is not in between 470um and 591um.
* Patients who have received lacrimal duct procedure within the last 3 months or who have plans to have it.
* pregnant or nursing women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-09-13 (Actual)

PRIMARY OUTCOMES:
Corneal staining test | (12-week-point)
  The degree of staining of the cornea after blue fluorescein staining under the light of cobalt blue using a yellow filter was evaluated according to the Oxford grading system (0 to 5, the higher the worse)
Conjunctival staining test | (12-week-point)
  The conjunctiva was divided into 6 areas and evaluated after the same staining method according to the Oxford grading system (0 to 3, the higher the worse)
Ocular surface disease index (OSDI) | (12-week-point)
  The ocular surface was assessed using OSDI scoring questionnaire (0 to 100, the higher the worse)
Compliance check | (12-week-point)
  Compliance of the drug administration has been check through the subject's self description (0 to 100, the higher the better)

SECONDARY OUTCOMES:
Corneal staining test | (4-week-point)
  The degree of staining of the cornea after blue fluorescein staining under the light of cobalt blue using a yellow filter was evaluated according to the Oxford grading system(0 to 5, the higher the worse)
Conjunctival staining test | (4-week-point)
  The conjunctiva was divided into 6 areas and evaluated after the same staining method according to the Oxford grading system (0 to 3, the higher the worse)
Ocular surface disease indext (OSDI) | (4-week-point)
  The ocular surface was assessed using OSDI scoring questionnaire(0 to 100, the higher the worse)
IOP (intraocular pressure) | (4- / 12-week-point)
  IOP was measured using Goldmann applanation tonometry and measured in mmHg. (numerical)
Tear break up time (TBUT) | (4- / 12-week-point)
  The time taken from the last blink to the appearance of a black spot on the cornea after fluorescein dye staining. (second, numerical)
Limbal and bulbar hyperemia | (4- / 12-week-point)
  The conjunctival hyperemia was assessed using Efron grading scales (0 to 4, the higher the worse)

CONTACTS AND LOCATIONS:
Overall Officials: Seungsoo Rho, MD, PhD, Principal Investigator — CHA Bundang Medical Center
Locations (1):
- CHA University Bundang Medical Center, Seongnam, Bundang-gu, South Korea